CLINICAL TRIAL: NCT03550911
Title: Constitution Of A Biological Collection From Samples From The Gut Microbiota In Patients Having A Bone Or Joint Infection Treated By A Suppressive Subcutaneous Antibiotherapy With Betalactamine (CARBAMICROBIOTA)
Brief Title: Biological Collection From Samples From The Gut Microbiota In Patients Having A Bone Or Joint Infection Treated By A Suppressive Subcutaneous Antibiotherapy With Betalactamine (CARBAMICROBIOTA)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0014
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Bone Infection; Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological collection from samples from the GUT microbiota in patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine. No analysis will be done for instance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biological Collection From Samples From The Gut Microbiota — The aim of this study is just to constitute a biological collection from samples from the Gut microbiota in patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine. No analysis will be done for instance.

SUMMARY:
Optimal surgical therapy (debridement in chronic osteomyelitis; device exchange in patients with chronic prosthetic joint infection (PJI)) could be sometimes non-feasible, especially in the elderly population. Therefore, a medical therapy with oral prolonged suppressive antibiotic therapy (PSAT) seems to be an option to prevent recurrence and prosthesis loosening. Unfortunately, some patients are infected with resistant pathogens for which oral antibiotics are not suitable. Subcutaneous (SC) administration of injectable intravenous antibiotics as prolonged suppressive antibiotic therapy could be a convenient way to limit catheter-related complications and facilitate ambulatory care.

However, there are few data concerning the development of resistance under subcutaneous prolonged treatment with betalactamine.

The aim of this study is just to constitute a biological collection from samples from the Gut microbiota in patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine. Later analysis will be led on those samples to detect the acquisition of resistance or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a bone or joint infection
* Patients treated by a suppressive subcutaneous antibiotherapy with betalactamine

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Biological Collection From Samples From The Gut Microbiota | 1 day
  The aim of this study is just to constitute a biological collection from samples from the Gut microbiota in patients having a bone or joint infection treated by a suppressive subcutaneous antibiotherapy with betalactamine.
  No analysis will be done for instance.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des infections ostéo-articulaires de Lyon - Hôpital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No